CLINICAL TRIAL: NCT00238537
Title: Echoplanar Imaging Thrombolysis Evaluation Trial (EPITHET) in Acute Stroke
Brief Title: Echoplanar Imaging Thrombolysis Evaluation Trial (EPITHET)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melbourne Health (Other)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 145671; TGA Trial Number: 1999/271; Enterprise ID: 15314
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2009-05

CONDITIONS: Stroke
Keywords: Stroke; Thrombolysis; MRI; Echoplanar; Penumbra
MeSH Terms: conditions — Stroke | interventions — PLAT protein, human

INTERVENTIONS:
Drug: Alteplase t-PA

SUMMARY:
To determine whether the extent of the ischemic penumbra apparent on perfusion-diffusion MRI can be used to identify patients who would respond positively and safely to tissue plasminogen activator (tPA) beyond 3 hours post-stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present:
* with acute hemispheric stroke within 3-6 hours of onset,
* have at least moderate limb weakness,
* a National Institute of Health Stroke Scale (NIHSS) score > 4,
* had a pre-stroke modified Rankin Scale (MRS) score of 0 - 2
* and who are able to undergo CT and MRI, are eligible for this study.

Exclusion Criteria:

* Females who are pregnant or breast-feeding,
* persons who have CT-verified hemorrhagic stroke, major ischemia ( > 33% of the middle cerebral artery (MCA) territory infarcted), subarachnoid hemorrhage, arteriovenous malformation, aneurysm, intracranial neoplasm that is terminal or poses a risk of hemorrhage ,
* are comatose or severely obtunded with fixed eye deviation and complete hemiplegia,
* have had another stroke within the past 6 weeks,
* have had a seizure prior to the administration of the study drug,
* have active peptic ulceration, bleeding diatheses, previous intracerebral hemorrhage,
* blood pressure > 185/110,
* major surgery or trauma within the past 30 days, or any other contraindications to tPA
* have a presumed septic embolus or a myocardial infarction within the past 30 days
* blood glucose values are < 2.8 or > 22.0 mmol/L,
* pacemakers, aneurysm clips, implanted devices, claustrophobia, or any other contraindications to MRI,
* decreased consciousness,
* rapid clinical improvement,
* confounding neurological condition (e.g. dementia),
* any other life-threatening illness, or who are participating in another clinical trial, will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2001-08; Study Completion 2007-04

PRIMARY OUTCOMES:
Primary Hypothesis - lesion growth
In patients with penumbra, there will be attenuation of lesion growth (outcome T2 lesion volume - acute DWI volume ) with tPA.

SECONDARY OUTCOMES:
Secondary Hypotheses
In the non-penumbral group, lesion growth will be lower and will not be attenuated by tPA.
Favourable functional outcome (mRS 0-2) will be more likely in patients with penumbra receiving tPA.
That the proportion of patients achieving good neurological outcome (an 8 point improvement in NIH-SS or outcome NIH-SS of 0, 1) will be greater in those patients with a penumbra receiving tPA.
Symptomatic hemorrhagic transformation (sICH) will be predicted by the size of the baseline DWI volume in those patients receiving tPA.
Reperfusion (greater than 90% PWI lesion reduction, or recanalisation on MRA, between the acute and sub-acute interval), will be increased (in patients with penumbra) receiving tPA.
In patients with malignant mismatch (Definition DWI 100ml or more and / or PWI 100ml or more) there will be unfavourable clinical outcome (even if there is attenuation of growth).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Davis, MD FRCP FRACP, Study Chair — Melbourne Health; Geoffrey Donnan, MD FRACP, Study Chair — National Stroke Research Institute, Australia
Locations (14):
- Australia (10):
  - Hunter New England Area Health Service, Newcastle, New South Wales
  - Royal Brisbane Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Center, Adelaide, South Australia
  - Royal Melbourne Hospital, Melbourne, Victoria
  - St Vincents Hospital, Melbourne, Victoria
  - Austin Hospital, Melbourne, Victoria
  - Box Hill Hospital, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Cliniques Universitaires St Luc, Brussels, Belgium
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
- Southern General Hospital, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Derived] Ogata T, Christensen S, Nagakane Y, Ma H, Campbell BC, Churilov L, Lansberg MG, Straka M, De Silva DA, Mlynash M, Bammer R, Olivot JM, Desmond PM, Albers GW, Davis SM, Donnan GA; EPITHET and DEFUSE Investigators. The effects of alteplase 3 to 6 hours after stroke in the EPITHET-DEFUSE combined dataset: post hoc case-control study. Stroke. 2013 Jan;44(1):87-93. doi: 10.1161/STROKEAHA.112.668301. Epub 2012 Dec 18. PMID 23250996
- [Derived] Mlynash M, Lansberg MG, De Silva DA, Lee J, Christensen S, Straka M, Campbell BC, Bammer R, Olivot JM, Desmond P, Donnan GA, Davis SM, Albers GW; DEFUSE-EPITHET Investigators. Refining the definition of the malignant profile: insights from the DEFUSE-EPITHET pooled data set. Stroke. 2011 May;42(5):1270-5. doi: 10.1161/STROKEAHA.110.601609. Epub 2011 Apr 7. PMID 21474799
- [Derived] Davis SM, Donnan GA, Parsons MW, Levi C, Butcher KS, Peeters A, Barber PA, Bladin C, De Silva DA, Byrnes G, Chalk JB, Fink JN, Kimber TE, Schultz D, Hand PJ, Frayne J, Hankey G, Muir K, Gerraty R, Tress BM, Desmond PM; EPITHET investigators. Effects of alteplase beyond 3 h after stroke in the Echoplanar Imaging Thrombolytic Evaluation Trial (EPITHET): a placebo-controlled randomised trial. Lancet Neurol. 2008 Apr;7(4):299-309. doi: 10.1016/S1474-4422(08)70044-9. Epub 2008 Feb 28. PMID 18296121